CLINICAL TRIAL: NCT06625151
Title: Perfectionism and Daily Stress, Coping, and Well-Being: Testing an Explanatory Feedback Intervention
Brief Title: Perfectionism and Daily Coping and Emotion Regulation Processes: A Trial of Two Explanatory Feedback Interventions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, David Dunkley, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fund #256468; SSHRC 435-2021-0581 (Other Grant/Funding Number: Social Sciences and Humanities Research Council of Canada)
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Perfectionism; Psychological Well-being; University Students
Keywords: Perfectionism; Stress; Coping; Emotion Regulation; Mood; Daily Diary; Feedback Intervention
MeSH Terms: conditions — Psychological Well-Being; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: The four conditions will be: (a) waitlist control condition, (b) PCPM-EFI, (c) PERPM-EFI, and (d) PCPM-EFI plus PERPM-EFI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Wait-list Control (No Intervention): After all the final outcome measures have been completed at T3 (two weeks after Time 2), participants will be offered the PCPM-EFI and PERPM-EFI.
- PCPM-EFI (Experimental): At Time 2 (two weeks after baseline), participants will receive the PCPM-EFI. Participants in the PCPM-EFI condition will be offered the PERPM-EFI after all assessments have been completed at Time 3.
  Interventions: Behavioral: Perfectionism and Coping Processes Model - Explanatory Feedback Intervention (PCPM-EFI)
- PERPM-EFI (Experimental): At Time 2 (two weeks after baseline), participants will receive the PERPM-EFI. Participants in the PERPM-EFI condition will be offered the PCPM-EFI after all assessments have been completed at Time 3.
  Interventions: Behavioral: Perfectionism and Emotion Regulation Processes Model - Explanatory Feedback Intervention (PERPM-EFI)
- PCPM-EFI plus PERPM-EFI (Experimental): At Time 2 (two weeks after baseline), participants will receive the PCPM-EFI plus the PERPM-EFI.
  Interventions: Behavioral: Perfectionism and Coping Processes Model - Explanatory Feedback Intervention (PCPM-EFI); Behavioral: Perfectionism and Emotion Regulation Processes Model - Explanatory Feedback Intervention (PERPM-EFI)

INTERVENTIONS:
Behavioral: Perfectionism and Coping Processes Model - Explanatory Feedback Intervention (PCPM-EFI) — The PCPM-EFI provides individualized explanatory feedback of daily diary data demonstrating how stress and coping processes for each participant trigger and maintain their negative and positive mood. The feedback consists of five separate modules: (a) how changes in perceived criticism, self-blame, perceived control, avoidant coping, and event stress are connected to increases negative affect; (b) how changes in perceived social support, positive reinterpretation, perceived control, avoidant coping, and problem-focused coping are linked to increases in positive affect; (c) how self-critical perfectionism and maladaptive stress and coping tendencies explain enduring mood problems; (d) how healthy striving, adaptive appraisal, and coping tendencies can identify personal strengths; and, most important, (e) what the person needs to do to manage and improve his or her mood.
  Arms: PCPM-EFI; PCPM-EFI plus PERPM-EFI
Behavioral: Perfectionism and Emotion Regulation Processes Model - Explanatory Feedback Intervention (PERPM-EFI) — The PERPM-EFI provides individualized explanatory feedback of daily diary data demonstrating how stress and emotion regulation processes for each participant trigger and maintain their negative and positive mood. The feedback consists of five separate modules: (a) how changes in event stress, mindfulness, self-compassion, experiential avoidance, and rumination are connected to increases in negative affect, (b) how changes in event stress, mindfulness, reappraisal, self-compassion, and experiential avoidance are linked to increases in positive affect, (c) how self-critical perfectionism and maladaptive stress and emotion regulation tendencies explain enduring mood problems, (d) how healthy striving, adaptive appraisal, and emotion regulation tendencies can identify personal strengths, and, most important, (e) what the person needs to do to manage and improve his or her mood.
  Arms: PCPM-EFI plus PERPM-EFI; PERPM-EFI

SUMMARY:
Over the past three decades, perfectionism has received increasing theoretical and empirical attention as a cognitive-personality factor that increases vulnerability to a wide range of psychological problems, including depression and anxiety. Although mediators and moderators of the link between perfectionism and well-being have been identified, the direct clinical utility of these findings has not been a focus. The Perfectionism and Coping Processes Model - Explanatory Feedback Intervention (PCPM-EFI) draws on previous findings and individually analyzes participant responses to perfectionism measures and online daily questionnaires of stress, coping, and mood over 7 days. The EFI provides an individualized slideshow presentation that is delivered in a single 45-60 minute session by a student research assistant to address how stress and coping patterns trigger and maintain negative affect and (lower) positive affect in the participant's daily life. A recent waitlist controlled feasibility trial compared the PCPM-EFI condition with a waitlist control condition over 4 weeks in 176 university students with higher SC perfectionism, with individualized feedback delivered one-on-one by student trainees in-person or remotely through videoconferencing. The feasibility of the individualized analyses of each participant's daily data was supported by identifying daily trigger patterns, maintenance tendencies, strengths, common triggers, and best targets for reducing negative mood and increasing positive mood across several stressors for each participant. Participant ratings indicated that the comprehensive feedback was coherent and functional. Participants in the EFI condition, compared to those in the control condition, reported increases in empowerment, coping self-efficacy, and problem-focused coping, as well as decreases in depressive and anxious symptoms. Between-group effect sizes were moderate-to-large. There were reliable improvements in empowerment and depressive symptoms for 56% and 36%, respectively, of participants in the EFI condition. These findings demonstrate the broad applicability, conceptual utility, and effectiveness of the PCPM-EFI for self-critical perfectionistic individuals. Given these promising findings, research is needed to examine the utility of customizing daily emotion regulation findings, and the complementary effects of providing meaningful feedback on well-being.

The present study will build on the promising findings of the PCPM-EFI by using a 7-day daily diary methodology to test a complementary EFI on perfectionism and emotion regulation processes (e.g., self-compassion, mindfulness, experiential avoidance, rumination, reappraisal) delivered online through videoconferencing in a sample of university students with higher self-critical perfectionism. Based on the Perfectionism and Emotion Regulation Processes Model (PERPM), the PERPM-EFI follows the same structure as the PCPM-EFI to provide individualized analyses drawn from previous findings. The results of a pilot study of 12 university students with higher SC perfectionism suggest that the PERPM-EFI is broadly applicable, conceptually useful, and effective. Specifically, despite the small sample size, participants reported increases in empowerment, mindfulness, self-compassion, and emotional self-awareness, as well as decreases in depressive and anxious symptoms. The present study will use a randomized control design to examine whether the PCPM-EFI plus PERPM-EFI can better improve well-being, relative to providing no feedback, the PERPM-EFI alone, or PCPM-EFI alone in the context of a 4-week longitudinal study with three time points in a sample of 180 university students. The four conditions will be: (a) waitlist control condition, (b) PCPM-EFI, (c) PERPM-EFI, and (d) PCPM-EFI plus PERPM-EFI. It is hypothesized that all three EFI conditions will yield better outcomes than the waitlist control condition. It is also hypothesized that the combined PCPM-EFI plus PERPM-EFI condition will be superior to the PCPM-EFI condition and PERPM-EFI condition on empowerment (primary outcome) and secondary symptom outcomes (i.e., depressive symptoms, anxious symptoms, negative affect, positive affect). It is also expected that participants in the PCPM-EFI plus PERPM-EFI condition and PCPM-EFI condition will exhibit larger increases in coping self-efficacy and problem-focused coping than participants in the PERPM-EFI condition. On the other hand, it is hypothesized that participants in the PCPM-EFI plus PERPM-EFI condition and PERPM-EFI condition will exhibit larger increases in self-compassion, mindfulness, and emotional self-awareness than participants in the PCPM-EFI condition. If the feedback interventions are shown to be efficacious, the interventions could be offered to universities, work places, clinical settings, and other organizations.

DETAILED DESCRIPTION:
1. Rationale for Study. Over the past three decades, perfectionism has received increasing theoretical and empirical attention as a cognitive-personality factor that increases vulnerability to several psychological problems, including depression and anxiety. In Canada, the United States, and the United Kingdom, young adults are experiencing higher levels of depression, anxiety, and suicide ideation as well as significantly higher levels of self-critical perfectionism than a decade ago. Although the self-criticism (SC) dimension of perfectionism has been consistently associated with lower well-being, little longitudinal research has examined the mechanisms through which SC is related to well-being over time.

1.a. Perfectionism Dimensions and Daily Stress Reactivity and Coping (In)effectiveness.

Previous longitudinal studies of university students, community adults, and depressed patients have used 7-day and 14-day daily diary designs to obtain several assessments of appraisals, coping, and affect for each individual in the individual's natural everyday environments. Based on the Perfectionism Coping Processes Model (PCPM), multilevel structural equation modeling (MSEM)/SEM between-persons results have demonstrated that SC perfectionists maintain lower well-being (e.g., negative affect, lower positive affect) over time because these individuals have a tendency to: (a) generate daily stress for themselves by magnifying the negative aspects of events such that mundane difficulties can be interpreted as threatening stressors; (b) engage in avoidant coping, which stems from helplessness thinking that the individual is unable to cope with stressors to the individual's own and others' satisfaction; and (c) perceive that others are unwilling or unavailable to help the individual in times of stress, and thereby lack an important resource (i.e., perceived social support) to make stressors seem less overwhelming. On the other hand, the adaptive potential of PS has been exhibited by an indirect relation with positive affect through maintenance of higher daily problem-focused coping when individuals with higher PS are not depressed. MSEM within-person results have shown that several distinct appraisals (e.g., event stress) and coping strategies (e.g., avoidant coping) commonly operate together across many different stressors when the typical individual experiences daily increases in negative affect and drops in positive affect. In parallel, constructive social (e.g., perceived social support) and self (e.g., perceived control) appraisals and engagement coping strategies (e.g., positive reinterpretation, problem-focused coping) commonly facilitate one another, which is linked to within-person increases in daily positive affect for the typical individual.

1.b. Perfectionism Dimensions and Daily Emotion (Dys)regulation. Given the pervasive and enduring stress management problems that generate persistent distress for perfectionistic individuals, it is important to better understand how certain emotion regulation strategies might make emotional reactions worse or serve a protective role. A recent SSHRC-funded study extends this previous research by using 14-day daily diaries and MSEM/multilevel modeling to examine the impact of SC and PS dimensions of perfectionism on emotion regulation (e.g., mindfulness, self-compassion, experiential avoidance, rumination) and well-being in a sample of 154 community adults over two years. Based on the Perfectionism and Emotion Regulation Processes Model (PERPM), MSEM between-persons results demonstrated that SC perfectionism maintains higher negative affect and lower positive affect over 14 days because these individuals have a tendency to generate daily stress for themselves and engage in experiential avoidance and rumination, and tend less to engage in mindfulness, self-compassion, and reappraisal. Within-person mediation results showed that, when the typical individual perceives more stress than usual, the individual responds with less mindfulness, self-compassion, and reappraisal than usual, and engages in more experiential avoidance and rumination than usual, and this was connected to decreases in daily well-being. Further, multilevel modeling results demonstrated that individuals with higher SC perfectionism, relative to those with lower SC, experience stronger within-person decreases in well-being (e.g., higher negative affect, lower positive affect) when the individual reports more stress than usual, and less self-compassion and mindfulness than usual.

1. c. Feedback Interventions for Perfectionists. Although mediators and moderators of the link between perfectionism and well-being have been identified, the direct clinical utility of these findings has not been a focus. Few studies have involved participants in a role beyond the completion of study questionnaires/diaries. An exception was a study in which a total of 60 young adults assessed to be maladaptive perfectionists were randomized to a control group or a single-session feedback intervention in which the participant's perfectionism results were discussed. Findings revealed that providing feedback to maladaptive perfectionists about the individual's perfectionism reduced self-reported global symptomatic distress as well as emotional reactivity. Although the findings suggest that a brief, individualized feedback intervention is effective, one important limitation of extant studies employing feedback interventions is that the feedback did not describe the actions to be taken to make change. According to feedback intervention theory and the model of actionable feedback, feedback will have an optimal effect on performance when information is focused on helping the recipient see how his/her behaviour should change to improve functioning. This entails customizability of feedback that engages the individual with his/her own data, making him/her an active participant in the sense-making process, rather than a passive recipient of information.

   The Perfectionism and Coping Processes Model - Explanatory Feedback Intervention (PCPM-EFI) draws on previous findings and analyzes participant responses to perfectionism measures and online daily questionnaires of stress, coping, and mood over 7 days. The PCPM-EFI provides an individualized slideshow presentation that is delivered in a single 45-60 minute session by a student research assistant to answer five questions about the participant's perfectionism and daily stress, coping, and affect patterns. Question 1 ("What increases the participant's negative mood?") is addressed by contrasting scores from two days with a path diagram to demonstrate to the individual that, when the individual perceives more criticism, engages in more self-blame, and/or perceives less control than usual, the individual uses more avoidant coping and/or experiences higher event stress than usual, and this is connected to daily increases in negative affect. Question 2 ("What increases the participant's positive mood?") is addressed by contrasting scores from two days with a path diagram to show to the individual that, when the individual perceives more support from others, uses more positive reinterpretation, and/or perceives more control than usual, the individual engages in more problem-focused coping than usual, and this is connected to daily increases in positive affect. Question 3 ("What's keeping the participant stuck?") is addressed by showing the individual how higher levels of SC maintained higher negative affect and lower positive affect averaged over seven days because of selected higher disengagement tendencies (e.g., stress, avoidant coping, perceived criticism, self-blame) and selected lower engagement tendencies (e.g., perceived social support, positive reinterpretation, perceived control, problem-focused coping). Question 4 ("What are the participant's strengths?") is addressed by highlighting strengths to the individual, including healthy striving (i.e., PS without SC), selected lower disengagement tendencies, and selected higher engagement tendencies averaged over seven days. Most important, Question 5 ("What can the participant do to improve the participant's mood?") is addressed with a summary slide to show what the person needs to do to manage and improve the individual's mood. A given mechanism is designated as a "best target" when it is keeping the individual stuck and daily changes are connected to improvements in at least one other mechanism and mood.

   The investigators recently completed a waitlist controlled feasibility trial comparing the PCPM-EFI condition with a waitlist control condition over 4 weeks in 176 university students with higher SC perfectionism, with individualized feedback delivered one-on-one by student trainees in-person or remotely through videoconferencing. The feasibility of the individualized analyses of each participant's daily data was supported by identifying daily trigger patterns, maintenance tendencies, strengths, common triggers, and best targets for reducing negative mood and increasing positive mood across several stressors for each participant. Participant ratings indicated that the comprehensive feedback was coherent and functional. Participants in the EFI condition, compared to those in the control condition, reported increases in empowerment, coping self-efficacy, and problem-focused coping, as well as decreases in depressive and anxious symptoms. Between-group effect sizes were moderate-to-large. There were reliable improvements in empowerment and depressive symptoms for 56% and 36%, respectively, of participants in the EFI condition. These findings demonstrate the broad applicability, conceptual utility, and effectiveness of the PCPM-EFI for self-critical perfectionistic individuals. Given these promising findings, research is needed to examine the utility of customizing daily emotion regulation findings, and the complementary effects of providing meaningful feedback on well-being.
2. The Present Study. The present SSHRC-funded study will build on the promising findings of the PCPM-EFI by using a 7-day daily diary methodology to test a complementary EFI on perfectionism and emotion regulation processes (e.g., self-compassion, mindfulness, experiential avoidance, rumination, reappraisal) delivered online through videoconferencing in a sample of university students with higher self-critical perfectionism. Based on the Perfectionism and Emotion Regulation Processes Model (PERPM), the PERPM-EFI follows the same structure as the PCPM-EFI to provide individualized analyses drawn from previous findings as well as findings from a current SSHRC-funded study. The results of a pilot study of 12 university students with higher SC perfectionism suggest that the PERPM-EFI is broadly applicable, conceptually useful, and effective. Specifically, despite the small sample size, participants reported increases in empowerment, mindfulness, self-compassion, and emotional self-awareness, as well as decreases in depressive and anxious symptoms. The present study will use a randomized control design to examine whether the PCPM-EFI plus PERPM-EFI can better improve well-being, relative to providing no feedback, the PERPM-EFI alone, or PCPM-EFI alone in the context of a 4-week longitudinal study with three time points in a sample of 180 university students. The four conditions will be: (a) waitlist control condition, (b) PCPM-EFI, (c) PERPM-EFI, and (d) PCPM-EFI plus PERPM-EFI.

   Based on theory and previous findings, it is expected that the EFIs will demonstrate three central features of the PCPM and PERPM as viable models of change (Hayes, Hofmann, and Ciarrochi, 2020). Hypothesis 1 will examine the feasibility of the individualized analyses of each participant's daily questionnaire data to show that the PCPM-EFI and PERPM-EFI are broadly applicable across a wide array of stressors for most participants in predictable, empirical ways. For each participant, it is expected that several appraisal, coping, emotion regulation, and affect scores will change together on a daily basis in a manner consistent with the Disengagement Trigger Patterns (Hypothesis 1a) and Engagement Trigger Patterns (Hypothesis 1b) described above. It is also expected that higher/lower levels of aggregated daily disengagement/engagement variables will differentiate each SC perfectionistic participant from the average person to fit the Explanatory Conceptualizations described above (Hypothesis 1c). It is also anticipated that many participants will exhibit some higher engagement and/or lower disengagement tendencies to support a Resilience Conceptualization (Hypothesis 1d), consistent with previous findings demonstrating the heterogeneity of perfectionism. Most important, it is also expected that for most participants there will be at least one disengagement or engagement variable that is both a maintenance tendency and a common trigger for the Best Target Selection for each of the PCPM-EFI and PERPM-EFI (Hypothesis 1e).

   Hypothesis 2 addresses the conceptual utility feasibility of the PCPM-EFI and PERPM-EFI steps, derived from the individualized outputs of each participant's daily diary data. Participant ratings will indicate that the participant (strongly) agrees that the comprehensive feedback of the EFI steps, as delivered by student research assistants, helps the participant understand and make sense of the individual's mood and is functional in helping the participant understand how to improve the individual's mood.

   Finally, Hypothesis 3 is that participants in the experimental conditions, compared to those in the control condition, will report primarily increases in empowerment (i.e., being better informed, improved acceptance of problems, increased optimism and control over the future, enhanced self-esteem). Empowerment is the primary outcome because the EFI steps predominantly function to make complex processes seem less overwhelming and more manageable to the individual by showing that situations unfold in expected ways and helping understand how problems are maintained, before the final step of selecting mechanisms for improving mood. It is hypothesized that all three EFI conditions will yield better outcomes than the waitlist control condition. It is also expected that the combined PCPM-EFI plus PERPM-EFI condition will be superior to the PCPM-EFI condition and PERPM-EFI condition on empowerment (primary outcome) and secondary symptom outcomes (i.e., depressive symptoms, anxious symptoms, negative affect, positive affect). It is also expected that participants in the PCPM-EFI plus PERPM-EFI condition and PCPM-EFI condition will exhibit larger increases in coping self-efficacy and problem-focused coping than participants in the PERPM-EFI condition. On the other hand, it is hypothesized that participants in the PCPM-EFI plus PERPM-EFI condition and PERPM-EFI condition will exhibit larger increases in self-compassion, mindfulness, and emotional self-awareness than participants in the PCPM-EFI condition. Reductions in SC perfectionism measures are not expected because the EFI does not directly target perfectionism itself and existing RCT data show that one session is insufficient for reducing perfectionism.
3. Research Plan.

3.a. Participants. Participants will be students at McGill University, including English- and French-speaking men and women between the ages of 18-65. Advertisements in student newspapers and bulletins placed around the McGill University campus and online advertisements will recruit university students. Individuals potentially interested in participating will be sent a link to complete the screening consent form online through Qualtrics. If a potential participant decides to take part in this study, the individual will be asked to complete the screening questionnaire as well as perfectionism and current mood questionnaires online in a 5-10 minute session to determine whether the individual qualifies to participate in the study.

3.b. Procedure. Participants who meet prescreening criteria will be randomly assigned to one of four conditions using the randomization function in Excel to ensure the right amount in each condition at the end of the study. At Time 1, participants will complete an online package of baseline measures at home to assess personality (e.g., perfectionism) and well-being (i.e., depression, anxiety, negative affect, positive affect). Next, participants will complete the online daily questionnaires once a day for seven consecutive days. At Time 2 (two weeks after baseline), all participants will complete the brief perfectionism and well-being measures online. The participants in the explanatory feedback conditions will receive personalized feedback about the individual's baseline questionnaire and daily diary results. Participants in the three different explanatory feedback conditions will receive either (a) the PCPM-EFI in a 45-60 minute session, (b) the PERPM-EFI in a 45-60 minute session, or (c) the PCPM-EFI and PERP-EFI in a combined 90-120 minute session. During this feedback session, participants will also be asked to provide feedback on the feedback intervention itself by completing questionnaires and providing verbal feedback. Selected outcome measures (5-10 minutes) will be completed immediately after the intervention. At Time 3 (two weeks after Time 2), participants will complete online the brief perfectionism and well-being measures.

After all assessments have been completed at Time 3, the participants in the waitlist control condition will be offered the PCPM-EFI and PERPM-EFI (90-120 minutes), the participants in the PCPM-EFI condition will be offered the PERPM-EFI (45-60 minutes), and the participants in the PERPM-EFI condition will be offered the PCPM-EFI (45-60 minutes) after all assessments have been completed at Time 3. Selected outcome measures (5-10 minutes) will be completed by the waitlist control, PCPM-EFI condition, and PERPM-EFI condition participants immediately after the intervention.

3.c. EFI Daily Diary Procedure. In this study, participants will complete seven daily diaries online. These portable electronic diaries have the capacity to present required items for questionnaires that are accessed by participants from a web link (http://qualtrics.com/), and to record, store, and export participant responses to statistical software (SPSS). Participants will be notified at 9:00pm to complete a daily self-report record at bedtime, any time between 9:00pm and 3:00am. It is also estimated that each recording will take participants approximately 14-18 minutes to complete. First, participants will rate on 5-point scales 26 items from the Positive and Negative Affect Scale (PANAS) to assess negative affect, positive affect, sadness, and hostility today, as in previous studies. Second, participants will rate on 9-point scales three items from the Test of Negative Social Interactions (TENSE) to indicate how frequently the participant had experienced different types of negative social interactions today, as in previous studies. Third, participants will rate on 7-point scales three appraisals of the most bothersome event or issue of today: unpleasantness, duration, and stressfulness. As in previous studies, these three appraisals will be combined to assess event stress. Two additional items will assess perceived control and perceived criticism. Fourth, participants will rate on 4-point scales how the participant coped with the individual's most bothersome issue today using seven selected 4-item scales from the situational version of the COPE to assess avoidant coping (behavioral disengagement, self-distraction, denial), problem-focused coping (active coping, planning), positive reinterpretation, and self-blame, consistent with previous studies. Fifth, participants will rate on 7-point scales three appraisals about the extent to which each of three social provisions were potentially available, wanted, and received in helping to handle the stressor today: reliable alliance, attachment, and guidance. As in previous studies, these three appraisals will be combined to assess perceived social support. Sixth, participants will report the extent to which the participant ruminated in response to the most bothersome event of the day by rating five modified items from the brooding subscale of the Ruminative Responses Scale (RRS). Seventh, participants will indicate the extent to which the participant engaged in emotion regulation behaviours with the most bothersome event or issue of the day by rating two items adapted from the Emotion Regulation Questionnaire (ERQ) to assess reappraisal and one additional modified item assessing reappraisal. Eighth, participants will indicate the extent to which the participant engaged in several experiential avoidance behaviours with the most bothersome event or issue of the day by rating eight items adapted from the Brief Experiential Avoidance Questionnaire (BEAQ). Ninth, participants will report the degree to which the participant used self-compassion (self-kindness vs self-judgment, common humanity vs isolation, mindfulness vs over-identification) skills in response to the most bothersome event of the day by rating 26 modified items from the Self-Compassion Scale (SCS). Finally, participants will report the degree to which the participant used mindfulness (observe, describe, acting with awareness, nonreactivity, nonjudgmental acceptance) skills in response to the most bothersome event of the day by rating 20 adapted items adapted from the Five Facet Mindfulness Questionnaire - Short Form (FFMQ-SF).

3.d. Data Analytics for the PCPM-EFI and PERPM-EFI. The Excel scoring program that was successfully used in the waitlist controlled feasibility trial of the PCPM-EFI was adapted to perform individualized analyses of the perfectionism and daily stress, emotion regulation (i.e., mindfulness, self-compassion, experiential avoidance, rumination), and affect questionnaire responses, based on recent PERPM findings in a sample of 154 community adults. The PCPM-EFI script manual that was successfully used to deliver the individualized results to participants in the waitlist controlled trial of the PCPM-EFI was adapted to develop the PERPM-EFI script manual to deliver the individualized PERPM results to participants. The PERPM-EFI addresses the same five within-person and between-persons questions of interest as the PCPM-EFI: (i) What increases negative mood?, (ii) What increases positive mood?, (iii) What maintains negative mood?, (iv) What maintains positive mood?, and (v) What needs to be done to improve mood?.

3.e. EFI Delivery. All participants will receive the feedback remotely through Zoom. The feedback intervention will be scheduled for one meeting per participant that lasts 45-60 minutes (the PCPM-EFI plus PERP-EFI session lasts 90-120 minutes). The meeting will be one-on-one, meaning that in each session, one research assistant will deliver feedback to one participant. The PCPM-EFI and PERPM-EFI are manualized and administered following a detailed script. Participants will also receive by e-mail a PDF of the graphical summaries of the individual's personalized feedback for the individual's own reference. Feedback sessions will be audio and visual recorded through Zoom. The audio plus visual recording will be deleted and the audio only recording will be downloaded from Zoom. The audiotape will be used for the purposes of providing feedback to the research assistants about the individual's delivery of the feedback intervention, as well as for reviewing participants' reactions to the feedback intervention.

3.f. EFI Training. The student research assistants will undergo 10 hours of feedback intervention training. Under the supervision and tutelage of the primary investigator, who is a licensed psychologist, the research assistants will practice administering feedback using the PCPM-EFI and PERPM-EFI protocols and role plays based on case examples from previous studies. If necessary, the research assistants will complete additional role plays until procedural uniformity is established. Differences will be measured by comparing participants' usability and acceptability ratings between feedback providers.

3.g. Conceptual Utility Questionnaire. Participants will be asked to rate two to three statements on the perceived helpfulness of the explanatory feedback to make sense of, clarify, and understand EFI steps: Disengagement Trigger Patterns, Engagement Trigger Patterns, Explanatory Conceptualization, Resilience Conceptualization, and Best Target Selection. Participants will provide ratings on 5-point scales (from strongly disagree to strongly agree) immediately after receiving the feedback for each of the EFI steps. After the Best Target Selection, participants will rate three additional statements on the perceived function of the feedback to help improve the individual's mood.

4. Data analyses. Multilevel regression will be used to analyze the effects of feedback condition on the change processes (i.e., empowerment, coping self-efficacy, coping, self-compassion, mindfulness, emotional self-awareness) and symptom outcomes (i.e., depressive, anxious, stress). Multilevel modeling analyses will allow separate regression coefficients to be estimated for each patient's scores across time in order to examine the influence of feedback condition on each change process and well-being variable. Group and Time main effects, together with Group × Time interactions, will be examined in each model. Between-group post hoc significance tests will be conducted. Reliable change will also be used in order to determine the number of participants becoming more empowered (primary outcome) and the number of participants with mild depressive symptoms (i.e., BDI scores of 10 or more) having less depressive symptoms (secondary outcome) after undergoing each EFI condition. Reliable change will also be used to determine the number of participants exhibiting less anxious symptoms, less stress, more coping self-efficacy, more problem-focused coping, more self-compassion, more mindfulness, and more emotional self-awareness after undergoing each EFI condition.

5. Sample Size and Justification. Out of 200 student participants, it is expected that 180 students will successfully complete all of the study assessments (estimated attrition rate of 10%). Between-group effect sizes were moderate-to-large for empowerment (d = 0.89), coping self-efficacy (d = 0.59), problem-focused coping (d = 0.43), depressive symptoms (d = -0.68), and anxious symptoms (d = -0.46) for 176 participants in the previous study testing the effectiveness of the PCPM-EFI. These anticipated effect sizes indicate that the expected sample of 45 participants per group will be sufficient to detect group differences in the present study. Recruitment and follow-up of participants will occur over the academic year (October 2024 to May 2026), and subsequent months/years will be spent analyzing and writing papers based on these findings. If the feedback interventions are shown to be efficacious, the interventions could be offered to universities, work places, clinical settings, and other organizations.

ELIGIBILITY:
Individuals potentially interested in participating will be prescreened for levels of SC perfectionism and negative and positive mood.

Inclusion Criteria:

* Included in the study will be students who score 0.5 standard deviation above the mean score on two or more of four brief [4- or 5-item] measures of SC perfectionism (DEQ self-criticism, FMPS concern over mistakes, HMPS socially prescribed perfectionism, and APS-R discrepancy) for previous student samples

Exclusion Criteria:

* Individuals who meet the criteria for a diagnosis of depression or anxiety disorders and who do not have concomitant mental health care will be excluded from the study.
* Participants will be excluded if they fail to complete any of the Time 1 measures, or seven days of the daily diary procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Patient Empowerment Scale - Adapted version (Dunkley et al., 2023; van Uden-Kraan et al., 2009) | Measure completed at Time 2 (two weeks after baseline) after all participants completed the Step 1 daily reporting procedure, and at Time 3 (two weeks after Time 2). Will also be administered immediately after feedback.
  20-item adapted measure of four empowering outcomes, including being better informed, improved acceptance of problems, increased optimism and control over the future, and enhanced self-esteem. All items have the format of a statement that begins with "Through my participation in the study, … ."

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI; Beck and Steer, 1987) | Measure completed at baseline, at Time 2 (two weeks after baseline), and at Time 3 (two weeks after Time 2).
  A 21-item measure of depression symptoms over the past week.
Depression, Anxiety, and Stress Scale-Short Form (DASS-21; Lovibond and Lovibond, 1995) | Measure completed at baseline, at Time 2 (two weeks after baseline), and at Time 3 (two weeks after Time 2).
  21-item measure of depressive, anxious, and stress symptoms over the past week.
Positive and Negative Affect Scale (PANAS; Watson et al., 1988) | Measure completed at baseline, at Time 2 (two weeks after baseline), and at Time 3 (two weeks after Time 2). Will also be administered immediately before and after feedback.
  A 26-item measure of negative affect, sadness, and positive affect over the past week.
Coping Self-Efficacy Scale (CSES; Chesney et al., 2006) | Measure completed at baseline, at Time 2 (two weeks after baseline), and at Time 3 (two weeks after Time 2). Will also be administered immediately after feedback.
  26-item measure assesses confidence in ability to perform behaviors important to adaptive coping, such as use problem-focused coping, stop unpleasant emotions and thoughts, and get support from friends and family.
COPE Inventory (Carver et al., 1989) | Measure completed at baseline, at Time 2 (two weeks after baseline), and at Time 3 (two weeks after Time 2).
  Seven selected 4-item scales from a time-limited version (i.e., during the past week) of the COPE Inventory (Carver et al., 1989) to assess avoidant coping (behavioral disengagement, self-distraction, denial), problem-focused coping (active coping, planning), positive reinterpretation, and self-blame, consistent with previous studies (Dunkley et al., 2000; Dunkley et al., 2017; Dunkley, Ma, et al., 2014; Dunkley et al., 2003).
Self-Compassion Scale (Neff, 2003) | Measure completed at baseline, at Time 2 (two weeks after baseline), and at Time 3 (two weeks after Time 2).
  A 26-item time-limited version of the SCS examines the extent to which participants engaged in self-compassion over the past week. Six subscales include self-kindness, self-judgment, common humanity, isolation, mindfulness, over-identification.
Five Facet Mindfulness Questionnaire (Baer et al., 2006) | Measure completed at baseline, at Time 2 (two weeks after baseline), and at Time 3 (two weeks after Time 2).
  39-item time-limited version of the FFMQ assesses the degree to which participants engage in mindfulness over the past week (observe, describe, acting with awareness, nonreactivity, nonjudgmental acceptance).
Ruminative Responses Scale (RRS; Treynor et al., 2003) | Measure completed at baseline, at Time 2 (two weeks after baseline), and at Time 3 (two weeks after Time 2).
  10-item time-limited version of the measure assesses the extent to which participants engaged in brooding or reflective pondering over the past week.
Brief Experiential Avoidance Questionnaire (BEAQ; Gámez et al., 2014) | Measure completed at baseline, at Time 2 (two weeks after baseline), and at Time 3 (two weeks after Time 2).
  15-item measure assesses the extent to which participants engage in experiential avoidance.
Emotional Self-Awareness Scale (ESAS; Kauer et al., 2012) | Measure completed at baseline, at Time 2 (two weeks after baseline), and at Time 3 (two weeks after Time 2).
  The 33-item ESAS has five subscales, including recognition, identification, communication, contextualization, and decision-making.
General, Academic, Social Hassles Scale for Students - Abbreviated version (GASHSS; Blankstein and Flett, 1993; Dunkley et al., 2003) | Measure completed at baseline, at Time 2 (two weeks after baseline), and at Time 3 (two weeks after Time 2).
  A 30-item measure of general, academic, and social hassles over the past week.
Brief Frost et al. (1990) Multidimensional Perfectionism Scale (FMPS) | Measure completed at baseline, at Time 2 (two weeks after baseline), and at Time 3 (two weeks after Time 2).
  A 10-item measure used to assess the personal standards subscale of PS perfectionism and the concerns over mistakes subscale of SC perfectionism.
Depressive Experiences Questionnaire - Short Form (DEQ; Rudich et al., 2008) | Measure completed at baseline, at Time 2 (two weeks after baseline), and at Time 3 (two weeks after Time 2).
  A 6-item measure of the self-criticism indicator of SC perfectionism.
Brief Slaney et al. (2001) Almost Perfect Scale-Revised (APS-R) | Measure completed at baseline, at Time 2 (two weeks after baseline), and at Time 3 (two weeks after Time 2).
  8-item measure assesses the high standards subscale of PS perfectionism and the discrepancy subscale of SC perfectionism.
Brief Hewitt and Flett (1991) Multidimensional Perfectionism Scale (HMPS) | Measure completed at baseline, at Time 2 (two weeks after baseline), and at Time 3 (two weeks after Time 2).
  A 10-item measure to assess the self-oriented perfectionism indicator of PS perfectionism and the socially prescribed perfectionism indicator of SC perfectionism.
Acceptance and Action Questionnaire (AAQ-II; Bond et al., 2011). | Measure completed at baseline, at Time 2 (two weeks after baseline), and at Time 3 (two weeks after Time 2).
  10-item measure assesses the extent to which participants engage in experiential avoidance.
Emotion Regulation Questionnaire (ERQ; Gross and John, 2003) | Measure completed at baseline, at Time 2 (two weeks after baseline), and at Time 3 (two weeks after Time 2).
  10-item scale measures the extent to which participants engage in reappraisal and expressive suppression.
Test of Negative Social Interactions (TENSE; Finch et al., 1999) | Measure completed at baseline, at Time 2 (two weeks after baseline), and at Time 3 (two weeks after Time 2).
  24-item time-limited measure assesses how frequently participants experienced different types of negative social interactions during the past week.
Social Provisions Scale (SPS; Cutrona and Russell, 1987). | Measure completed at baseline, at Time 2 (two weeks after baseline), and at Time 3 (two weeks after Time 2).
  12-item brief measure assesses the perceived availability of three social provisions: reliable alliance, attachment, and guidance.

CONTACTS AND LOCATIONS:
Overall Officials: David Dunkley, Ph.D., Principal Investigator — McGill University
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tobin R, Dunkley DM. Self-critical perfectionism and lower mindfulness and self-compassion predict anxious and depressive symptoms over two years. Behav Res Ther. 2021 Jan;136:103780. doi: 10.1016/j.brat.2020.103780. Epub 2020 Nov 23. PMID 33259957
- [Background] Moroz M, Dunkley DM. Self-critical perfectionism, experiential avoidance, and depressive and anxious symptoms over two years: A three-wave longitudinal study. Behav Res Ther. 2019 Jan;112:18-27. doi: 10.1016/j.brat.2018.11.006. Epub 2018 Nov 13. PMID 30466031
- [Background] Aldea MA, Rice KG, Gormley B, Rojas A. Telling perfectionists about their perfectionism: Effects of providing feedback on emotional reactivity and psychological symptoms. Behav Res Ther. 2010 Dec;48(12):1194-203. doi: 10.1016/j.brat.2010.09.003. Epub 2010 Sep 17. PMID 20933221
- [Background] Dunkley DM, Lewkowski M, Lee IA, Preacher KJ, Zuroff DC, Berg JL, Foley JE, Myhr G, Westreich R. Daily Stress, Coping, and Negative and Positive Affect in Depression: Complex Trigger and Maintenance Patterns. Behav Ther. 2017 May;48(3):349-365. doi: 10.1016/j.beth.2016.06.001. Epub 2016 Jun 9. PMID 28390498
- [Background] Dunkley DM, Zuroff DC, Blankstein KR. Self-critical perfectionism and daily affect: dispositional and situational influences on stress and coping. J Pers Soc Psychol. 2003 Jan;84(1):234-52. PMID 12518982
- [Background] Dunkley DM, Mandel T, Ma D. Perfectionism, neuroticism, and daily stress reactivity and coping effectiveness 6 months and 3 years later. J Couns Psychol. 2014 Oct;61(4):616-33. doi: 10.1037/cou0000036. Epub 2014 Aug 11. PMID 25111703
- [Background] Dunkley DM, Richard A, Tobin R, Saucier AM, Gossack A, Zuroff DC, Moskowitz DS, Foley JE, Russell JJ. Empowering self-critical perfectionistic students: A waitlist controlled feasibility trial of an explanatory feedback intervention on daily coping processes. J Couns Psychol. 2023 Oct;70(5):584-594. doi: 10.1037/cou0000691. Epub 2023 Jun 29. PMID 37384489
- [Background] Dunkley DM, Ma D, Lee IA, Preacher KJ, Zuroff DC. Advancing complex explanatory conceptualizations of daily negative and positive affect: trigger and maintenance coping action patterns. J Couns Psychol. 2014 Jan;61(1):93-109. doi: 10.1037/a0034673. PMID 24447060